CLINICAL TRIAL: NCT07323264
Title: SAS 1: Develop Ocular Disease (OSD) Diagnostic, Algorithms, and Management Protocols for Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Louis Tong (Other Government)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor-Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Organization: Singapore National Eye Centre (Other Government)
Other Study IDs: 2025-0126; 2025-0126 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2025-11-25; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye
Keywords: Cataract; EDOF; Monofocal IOL; Toric IOL; Post Lasik; High Corneal Astigmatism
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears Sample (Schirmers Test)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Post LVC with Dry Eye undergoing cataract surgery: Post LVC with Dry Eye undergoing cataract surgery
- High corneal Astigmatism with Dry Eye undergoing cataract surgery: High corneal Astigmatism with Dry Eye undergoing cataract surgery
- Dry eye with no other risk factor undergoing cataract surgery: Dry eye with no other risk factor undergoing cataract surgery
- Patient undergoing Cataract Surgery implanted with EDoF/ EDoF Toric IOL With Dry Eye: Patient undergoing Cataract Surgery implanted with EDoF/ EDoF Toric IOL With Dry Eye
- Patient undergoing Cataract Surgery implanted with Multifocal/ MultifocalToric IOL With Dry Eye: Patient undergoing Cataract Surgery implanted with Multifocal/ MultifocalToric IOL With Dry Eye
- Patient undergoing Cataract Surgery implanted with Toric IOL With Dry Eye: Patient undergoing Cataract Surgery implanted with Toric IOL With Dry Eye
- Patient undergoing Cataract Surgery implanted with Monofocal IOL With Dry Eye: Patient undergoing Cataract Surgery implanted with Monofocal IOL With Dry Eye
- Patient undergoing Cataract Surgery implanted with EDoF/ EDoF Toric IOL Without Dry Eye: Patient undergoing Cataract Surgery implanted with EDoF/ EDoF Toric IOL Without Dry Eye
- Patient undergoing Cataract Surgery implanted with Multifocal/ MultifocalToric IOL Without Dry Eye: Patient undergoing Cataract Surgery implanted with Multifocal/ MultifocalToric IOL Without Dry Eye
- Patient undergoing Cataract Surgery implanted with Toric IOL Without Dry Eye: Patient undergoing Cataract Surgery implanted with Toric IOL Without Dry Eye
- Patient undergoing Cataract Surgery implanted with Monofocal IOL Without Dry Eye: Patient undergoing Cataract Surgery implanted with Monofocal IOL Without Dry Eye

SUMMARY:
Patient: Tear film issues resulting in poor visual outcomes are a major cause of dissatisfaction after cataract surgery. There is no universal best preoperative algorithm for managing the ocular surface prior to surgery.

Industry: Recent advances in tear/cornea imaging and refractive cataract surgery such as multifocal intraocular lenses will be advantageous to patients only if tear film issues can be addressed.

Society: Cataract surgery is the most common ophthalmic surgery done in Singapore and worldwide. Improving vision by attending to tear film problems improves quality of life.

DETAILED DESCRIPTION:
Phase 1: Investigate the impact of ocular surface disease (OSD) on post-operative outcomes in cataract surgery.

Phase 1A: Longitudinal interventional parallel group study; small cohort to determine the impact of moderate dry eye for at-risk patient groups.

Phase 1B: Longitudinal interventional parallel group study; larger cohort of to compare outcomes based on different IOL types.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for dry eye (participant must meet at least 1 of the inclusion criteria below):

  1. Symptomatic for dry eye based on DEQ5 (>6) and [either TBUT less than 5 s or staining >grade 1 in any zone of the cornea]
  2. Either use of diquasfosol, cyclosporine eyedrops or tacrolimus eyedrops for dry eye disease in the last 2 weeks (and previously started for more than 2 months), OR current and visible lower punctal plugs in at least one eye

Inclusion criteria to fulfil all for controls (patients w/o dry eye):

1. DEQ5 <=6.
2. Staining < grade 1 in at least one corneal zone.
3. Not using diquasfosol, cyclosporine, tacrolimus in last 2 months.
4. No visible punctal plugs.

Exclusion Criteria:

* If there is another ocular condition which affects vision as much as cataract: active corneal stromal disease or scar or significant corneal endothelial disease
* Known diagnosis of active thyroid dysfunction, Sjogren disease and rheumatoid arthritis
* Intraocular surgery within the previous 6 months
* Laser-assisted in situ keratomileusis or pterygium surgery within the previous 3 months
* Central nervous system and hormonal drugs required within the last month and during the study
* Active ocular infection, inflamed chalazion, or presence of pterygium
* Glaucoma which requires topical anti-glaucoma medications
* Any need to wear contact lens during the study
* Having issues which make it difficult to follow up (eg., wheelchair, etc)
* Pregnant and breast-feeding woman

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient undergoing cataract surgery that met the study inclusion and exclusion
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | From pre-op to Post Operative 3 to 6 weeks
  Postoperative uncorrected visual acuity and repeatability of Biometry and Keratometry

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore